CLINICAL TRIAL: NCT00809458
Title: A Phase III Biomarker Study of Neoadjuvant Vitamin E in Patients With Locally Treatable Prostate Cancer Prior to Prostatectomy or Brachytherapy
Brief Title: Biomarker Study of Neoadjuvant Vitamin E in Patients With Locally Treatable Prostate Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low rate of accrual.
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INST 0808; NCI-2011-02662 (Registry Identifier: NCI Clinical Trials Reporting Program)
Record Dates: First submitted 2008-12-15; First posted 2008-12-17 (Estimated); Results first posted 2015-06-23 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Prostate Cancer
Keywords: Vitamin E; Prostate Cancer; Alpha-tocopherol (α-tocopherol)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Vitamin E; alpha-Tocopherol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Vitamin E) (Experimental): Vitamin E
  Interventions: Drug: Vitamin E
- Arm 2 (Placebo Comparator): Placebo (same vehicle as used for vitamin E)
  Interventions: Drug: Vitamin E

INTERVENTIONS:
Drug: Vitamin E — Patients will take one 400 IU tablet of vitamin E or a placebo daily. Patients will continue on this treatment from the time of randomization to the day before surgery or the brachytherapy procedure. This is expected to be between 4 to 6 weeks. The patient will continue with his regular medications. The vitamin E will be supplied by the clinical trial through the UNM CRTC pharmacy.
  Other Names: Alpha-tocopherol (α-tocopherol)

SUMMARY:
The purpose of this study is to find out if vitamin E can help treat prostate cancer. Vitamin E acts primarily as an anti-oxidant. By decreasing the oxidation in the cancer cell, the tumor cells may die. Vitamin E is a commonly used vitamin that has not been approved by the Food and Drug Administration for use in this type of cancer or for any known cancer. This study will test the hypothesis that vitamin E, in the setting of an oxidative stress such as smoking, can reduce prostate cancer related biomarkers in patients with localized prostate cancer in the neoadjuvant setting.

DETAILED DESCRIPTION:
- Prostate Cancer

Prostate cancer is the most common malignancy in American men. It was estimated that nearly 235,000 men in the United States would be diagnosed with prostate cancer and nearly 27,000 men would die. The treatment of localized prostate cancer includes surgery, radiation therapy, or watchful waiting. The relative benefits of these approaches is unclear and treatment choices are individualized and often patient driven. There is currently no proven benefit to receiving preoperative hormonal therapy for patients undergoing radical prostatectomy. As opposed to patients undergoing external beam radiation therapy, for patients undergoing brachytherapy pre treatment hormonal therapy is used in approximately 40% of patients. Thus, these patients offer a unique opportunity to test novel agents in the neoadjuvant setting.

- Vitamin E

The term vitamin E was introduced by Evans and Bishop to describe a dietary factor important for reproduction in rats. Natural vitamin E includes two groups of closely related fat-soluble compounds, the tocopherols and tocotrienols. Eight analogous compounds are widely distributed in nature. Rich, natural sources of vitamin E are edible plant oils. Distinct biological effects of different forms of vitamin E can be distinguished at a molecular level. Vitamin E is the major hydrophobic chain-breaking antioxidant that prevents the propagation of free radical reactions in the lipid components of membranes, vacuoles and plasma lipoproteins.

As an antioxidant, vitamin E acts in cell membranes where it prevents the propagation of free radical reactions. Non-radical oxidation products are formed by the reaction between alpha-tocopheryl radical and other free radicals, which are conjugated to glucuronic acid and excreted through the bile or urine. Vitamin E is transported in plasma lipoproteins.

Most studies of the safety of vitamin E supplementation have lasted for several months or less, so there is little evidence for the long-term safety of vitamin E supplementation. The Food and Nutrition Board of the Institute of Medicine has set an upper tolerable intake level (UL) for vitamin E at 1,000 mg (1,500 IU) for any form of supplementary alpha-tocopherol per day. Based for the most part on the result of animal studies, the Food and Nutrition Board decided that because vitamin E can act as an anticoagulant and may increase the risk of bleeding problems this is the highest dose unlikely to result in bleeding problems (http://dietary-supplements.info.nih.gov/factsheets/vitamin.asp).

The dose of vitamin E used in the Selenium and vitamin E prostate cancer prevention trial (the SELECT trial) was 400 IU per day and thus this is the dose chosen for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically or cytologically confirmed prostate cancer.
2. Patients must have localized prostate cancer and have decided to undergo a prostatectomy or brachytherapy.
3. Patient must not be taking supplemental vitamin E.
4. Age >18 years.
5. Life expectancy of greater than 6 months.
6. ECOG performance status =< 2.
7. Patients must have normal organ and marrow function as defined below:

   * leukocytes >= 3,000/mcL
   * absolute neutrophil count >=1,500/mcL
   * platelets >=100,000/mcL
   * total bilirubin within normal institutional limits
   * AST/ALT =< 2.5 X institutional upper limit of normal
   * creatinine =< 1.5 X normal institutional upper limit of normal
   * INR =<1.4
   * PTT =<1.4 X institutional upper limit of normal
8. Patients must have the ability to understand, and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have metastatic prostate cancer.
2. Patients may not be receiving any other investigational agents.
3. Patients with a known bleeding diathesis or patients on therapeutic anticoagulation. (This does not include the use of aspirin but refers to warfarin, heparin, or low molecular weight heparins).
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to vitamin E.
5. The patient may not receive a gonadotrophin release agonist (such as goserelin, or leuprolide), or an antiandrogen (such as bicalutamide, flutamide, or nilutamide) during the study.
6. Uncontrolled intercurrent illness that would limit compliance with study requirements.

   * Inclusion of Women and Minorities

     * Only men are eligible for this trial. Members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-09; Primary Completion 2010-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, M.D., Study Director — University of New Mexico Cancer Center; Richard Lauer, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico - Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org
- See also: UNM Cancer Center — http://www.cancer.unm.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at oncology clinics between December 2008 and April 2010. The study was terminated due to low accrual rate.
Pre-assignment Details: One subject suffered an unrelated bone fracture prior to study start, and another was determined to have metastatic disease. 71 participants were screened. 31 did not meet criteria; 25 refused study entry. 15 were enrolled
Groups:
- Arm 1 (Vitamin E): Vitamin E administration: one 400 IU tablet of vitamin E daily
- Arm 2 (Placebo): Placebo (same vehicle as used for vitamin E): one placebo tablet daily
Period: Overall Study
Arm/Group | Arm 1 (Vitamin E) | Arm 2 (Placebo)
Started | 9 | 6
Completed | 8 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Vitamin E) | Arm 2 (Placebo) | Total
Number analyzed (Participants) | 9 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 4 | 11
  >=65 years | 2 | 2 | 4
Age, Continuous [Median (Full Range); unit: years] | 60 [51 to 73] | 60.5 [52 to 66] | 60 [51 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 9 | 6 | 15
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Reduce Biomarkers of Prostate Cancer (PSA Blood Level)
Description: PSA levels will be measured as a sensitive marker of anti-androgenic activity that is a critical endpoint to be measured in this study. PSA blood levels will be determined at the initiation and completion of Vitamin E supplementation from blood obtained at these time points. A clinical reference laboratory will perform blood PSA analysis and will be compared with plasma cholesterol levels as a relative control.
Time Frame: 30 days
Population: This study was terminated early due to low accrual. No participants were analyzed for this outcome measure because the study was terminated. There are no data to report.
Arm/Group | Arm 1 (Vitamin E) | Arm 2 (Placebo)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Determine the Tolerability/Toxicity of a Short Course of Vitamin E in the Neoadjuvant Setting.
Description: 1. Cardiovascular Effects/ Thrombophlebitis
  2. Dermatologic Effects
  3. Gastrointestinal Effects (Gingival bleeding, and gastrointestinal irritations including: diarrhea, nausea, flatulence and stomach cramps)
  4. Hematologic Effects (Increased bleeding tendencies in vitamin K deficient patients; inhibition of prothrombin production
  5. Hepatic Effects (Vasculopathic hepatotoxicity and cholestasis)
  6. Neurologic Effects (Dizziness, headache, fatigue or weakness
  7. Ophthalmic Effects ( Blurred vision)
  8. Respiratory Effects (Pulmonary embolism)
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Arm 1 (Vitamin E) | Arm 2 (Placebo)
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Determine Concordance of the Biomarkers in This Setting
Description: The correlation between the ATQ level and the androgen receptor will be explored.
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | Arm 1 (Vitamin E) | Arm 2 (Placebo)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects were followed from the start of treatment until 30 days after prostatectomy or brachytherapy.
Arm/Group | Arm 1 (Vitamin E) | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 1/9 | 0/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Vitamin E) (N=9) | Arm 2 (N=6)
Hypotension (Low blood pressure) (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes